CLINICAL TRIAL: NCT02332317
Title: A Randomized, Controlled Phase III Study of Integrated, Specialized Palliative Rehabilitation for Patients With Newly Diagnosed Non-resectable Cancer.
Brief Title: Early, Integrated, Specialized Palliative Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vejle Hospital (Other)
Collaborators: Bispebjerg Hospital (Other); Danish Cancer Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pal-Rehab
Record Dates: First submitted 2014-12-30; First posted 2015-01-06 (Estimated); Last update posted 2021-06-01 (Actual); Status verified 2018-09

CONDITIONS: Advanced Cancer
Keywords: Advanced cancer; Early integration; Palliative rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control arm (No Intervention): 150 patients will receive standard oncology treatment.
- Intervention arm (Active Comparator): 150 patients will receive standard oncology treatment alongside a 12-week specialized palliative rehabilitation program
  Interventions: Behavioral: Palliative rehabilitation

INTERVENTIONS:
Behavioral: Palliative rehabilitation — 12-week individually customized, specialized palliative rehabilitation program
  Arms: Intervention arm

SUMMARY:
The purpose of this study is to identify whether patients with newly diagnosed advanced cancer benefit from a 12-week palliative rehabilitation program integrated with standard oncology treatment.

DETAILED DESCRIPTION:
300 patients with newly diagnosed advanced cancer are planned to be enrolled. They wil be randomized at a 1:1 ratio to standard oncology treatment or standard oncology treatment plus a 12-week individually customized palliative rehabilitation program.

The intervention takes place in a specialized palliative setting and is planned after an individual consultation with the patient and his relatives. It can be adjusted during the 12 weeks according to the patient's symptoms and needs. All or part of the palliative rehabilitation program is organized as weekly group sessions at the hospital. The group sessions consist of lectures and debates followed by physical training. Professionals involved in the group sessions are doctors, nurses, physiotherapists, psychologists, occupational therapists, social workers, dietitians, and a priest.

If needed, the patient and/or his relatives can also be offered individual sessions.

All contacts with the patients or his relatives during the 12 weeks are registered in order to document the intervention retrospectively.

The intervention is evaluated using questionnaires. All participants receive a questionnaire at baseline and after 6 and 12 weeks. The questionnaire consists of EORTC-QLQ-C30 (a validated questionnaire developed to assess the quality of life of cancer patients) and HADS (the validated Hospital Anxiety and Depression Scale). At baseline the questionnaire is extended with the question: "Which of the following problems/ symptoms do you need help with the most?". The patients can choose between 12 defined problems matching 12 of the scales of EORTC-QLQ-C30 or "none of the above". The answer given by the patient is labeled "The Primary Problem".

ELIGIBILITY:
Inclusion Criteria:

Participants must:

* be diagnosed with non-resectable cancer less than 8 weeks before inclusion. For patients with prostate cancer they must be refered to systemic oncology treatment for the first time less than 8 weeks before inclusion.
* be fit to receive standard oncology treatment and accepting treatment
* read and understand Danish
* sign informed consent

Exclusion Criteria:

* contact with a specialized palliative unit within the last year before inclusion
* unability to cooperate in the study
* missing informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Effect of the intervention on "The Primary Problem" chosen by the patient. | 6 and 12 weeks
  Comparing change from baseline to the weighed average of the 6 and 12-week follow-up of the scale in EORTC-QLQ-C30 that correlates to "The Primary Problem" of the patient (measured as area under the curve (AUC) of the change). If the patient has not chosen a "Primary Problem" the same measurement is done with the general health related quality of life scale.

SECONDARY OUTCOMES:
Effect of the intervention on all symptoms and problems present in the EORTC-QLQ-C30 Questionnaire | 6 and 12 weeks
  Comparing change from baseline to the weighed average of the 6 and 12 week follow-up of all the scales of EORTC-QLQ-C30 (measured as area under the curve (AUC) of the change).
Effect of the intervention on worries and symptoms of anxiety and depression | 6 and 12 weeks
  Comparing HADS-scores in the two arms
All cause mortality | 3 months after last data collection
  Comparing mortality in the two arms using Kaplan-Meier survival curve.
Economic consequences | 3 months after last data collection
  Comparing health related expenses in the two arms using register information about admissions to hospitals, visits with family doctors, emergency rooms etc.

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Jensen, Assoc. prof., Study Chair — Vejle Hospital
Locations (1):
- Department of Oncology, Vejle Hospital, Vejle, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nottelmann L, Groenvold M, Vejlgaard TB, Petersen MA, Jensen LH. Early, integrated palliative rehabilitation improves quality of life of patients with newly diagnosed advanced cancer: The Pal-Rehab randomized controlled trial. Palliat Med. 2021 Jul;35(7):1344-1355. doi: 10.1177/02692163211015574. Epub 2021 May 17. PMID 34000886
- [Derived] Nottelmann L, Groenvold M, Vejlgaard TB, Petersen MA, Jensen LH. A parallel-group randomized clinical trial of individually tailored, multidisciplinary, palliative rehabilitation for patients with newly diagnosed advanced cancer: the Pal-Rehab study protocol. BMC Cancer. 2017 Aug 23;17(1):560. doi: 10.1186/s12885-017-3558-0. PMID 28835218